CLINICAL TRIAL: NCT05969925
Title: Study of Some Biomarkers Of Heart Failure In Children Attending Pediatric Cardiology Department Of Assiut University Children Hospital
Brief Title: Biomarkers of Pediatric Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ahmed Ali Mahny (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Ahmed Ali Mahny, Specialist, Pediatric Hospital, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Ahmed Mahny
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: new biomarkers for heart failure — assess efficacy of new biomarkers for heart failure

SUMMARY:
Heart failure (HF) is a clinical syndrome where the heart is unable to pump the blood required to meet the metabolic demands of the body. Heart failure in children can result from a variety of structural or functional cardiac disorders with subsequent failure of the ventricles to fill with or eject blood

DETAILED DESCRIPTION:
Cardiac biomarkers are useful as diagnostic and prognostic tools, especially in patients with atypical signs and symptoms. High rate of complication in HF led to the search for suitable cardiac biomarker that diagnose heart failure as early as possible, predict outcome, reflect response to treatment and help in staging of heart failure and determine risk (6) . In pediatrics, biomarkers of heart failure are particularly important for the early identification and risk stratification of patients with systemic diseases and associated risk for early development of heart failure. Good biomarkers have the following characteristics: high sensitivity and specificity, the possibility of simultaneous processing of many samples, short analysis time, low cost, and good clinical applications, thus predicting the risk of heart failure and the associated prognosis as well as the adequacy of monitoring [7].

. Neutrophil gelatinase-associated lipocalin (NGAL) is a 25 kDa protein covalently bound to matrix metalloproteinase-9 which was first isolated from neutrophils. It belongs to the lipocalin family, NGAL has been found to be elevated in both plasma and urine in patients with HF.(8) NGAL also acts as a growth and differentiation factor in the renal epithelium [9].

ELIGIBILITY:
Inclusion Criteria Children from 1 month to 16 years old admitted to Assiut children University Hospital the Pediatric Cardiology unit with clinical manifestation of heart failure according to Ross classification either due to congenital or due to acquired heart disease will be enrolled in the study Exclusion Criteria Children with renal disease or failure, hepatic disease, pulmonary diseases will also excluded.

Ages: 1 Month to 16 Years | Sex: All
Age Groups: Child
Study Population: This study will be carried out in the children diagnosed with heart failure (HF) will be enrolled in this study. They will be choosen from those admitted at the Pediatric Cardiology Unit, Pediatric Department, Assiut University Children's Hospital in one year
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-02 (Estimated); Study Completion 2024-09-02 (Estimated)

PRIMARY OUTCOMES:
serum level of Neutrophil gelatinase-associated lipocalin in pediatric heart failure | one year
  accuarcy of serum level of Neutrophil gelatinase-associated lipocalin in heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Moahmmed, Dr., Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Watanabe K, Shih R. Update of Pediatric Heart Failure. Pediatr Clin North Am. 2020 Oct;67(5):889-901. doi: 10.1016/j.pcl.2020.06.004. Epub 2020 Aug 11. PMID 32888688